CLINICAL TRIAL: NCT02649426
Title: The "RADIANCE-HTN" Study. A Study of the ReCor Medical Paradise System in Clinical Hypertension
Brief Title: A Study of the ReCor Medical Paradise System in Clinical Hypertension
Acronym: RADIANCE-HTN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN 0777
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Vascular Diseases
Keywords: denervation; resistant hypertension; essential hypertension
MeSH Terms: conditions — Hypertension; Vascular Diseases; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound Renal Denervation (Experimental): Subjects in the TRIO or SOLO cohorts that are randomized to treatment, will receive renal denervation following a renal angiogram
  Interventions: Device: The Paradise® Renal Denervation Ultrasound System
- Sham Procedure (Sham Comparator): For subjects in TRIO or SOLO cohorts that randomize to the sham procedure, the diagnostic renal angiogram intervention will be considered the sham procedure.
  Interventions: Device: Sham Procedure

INTERVENTIONS:
Device: The Paradise® Renal Denervation Ultrasound System — Randomization will occur following the diagnostic renal angiogram. Blinded patients randomized to treatment will receive the renal denervation procedure using the Paradise System to deliver ultrasound energy to thermally ablate and disrupt the renal sympathetic nerves while sparing the renal arterial wall.
  Other Names: renal denervation
  Arms: Ultrasound Renal Denervation
Device: Sham Procedure — Randomization will occur following the diagnostic renal angiogram. For blinded patients randomized to control, the diagnostic renal angiogram will be considered the sham procedure.
  Other Names: renal angiogram
  Arms: Sham Procedure

SUMMARY:
RADIANCE-HTN is a randomized, double-blind, sham controlled, 2-cohort study (TRIO and SOLO) designed to demonstrate efficacy and document the safety of the Paradise Renal Denervation System in two distinct populations of hypertensive subjects.

DETAILED DESCRIPTION:
Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications will be included in the RADIANCE Solo cohort while subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications will be included in the RADIANCE Trio cohort. Prior to randomization, subjects will be hypertensive in the absence of hypertension medication (SOLO) or despite the presence of a stabilized, single pill, triple, fixed dose antihypertensive medication regimen (TRIO).

ELIGIBILITY:
TRIO and SOLO Inclusion Criteria:

* Appropriately signed and dated informed consent
* Age ≥18 and ≤75 years at time of consent
* Documented history of essential hypertension
* SOLO Cohort only: Either an average seated office BP < 180/110 mmHg at screening visit while on a stable regimen of 1 or 2 antihypertensive medications for at least 4 weeks prior to consent or an average seated office BP ≥ 140/90 mmHg <180/110 mmHg despite lifestyle measures on no antihypertensive medications
* TRIO Cohort only: Average seated office BP ≥ 140/90 mmHg at screening visit while on a stable regimen of at least 3 antihypertensive medications of different classes including a diuretic for at least 4 weeks prior to consent
* Documented daytime ABP ≥ 135/85 mmHg and < 170/105 mmHg after 4-week washout/run-in period (SOLO cohort) or after 4-week stabilization period (TRIO cohort)
* Suitable renal anatomy compatible with the renal denervation procedure and documented by renal CTA or MRA of good quality performed within one year prior to consent (a CTA or MRA will be obtained in patients without a recent (≤1 year) renal imaging)
* Able and willing to comply with all study procedures

Solo Exclusion Criteria:

* Renal artery anatomy on either side, ineligible for treatment including:

  * Main renal artery diameter < 4 mm and > 8 mm
  * Main renal artery length < 25 mm
  * A single functioning kidney
  * Presence of abnormal kidney (or secreting adrenal) tumors
  * Renal artery with aneurysm
  * Pre-existing renal stent or history of renal artery angioplasty
  * Prior renal denervation procedure
  * Fibromuscular disease of the renal arteries
  * Presence of renal artery stenosis of any origin ≥ 30%
  * Accessory arteries with diameter ≥ 2mm <4 mm and > 8 mm*
* Evidence of active infection within 7 days of procedure
* Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter
* Type I diabetes mellitus or uncontrolled Type II diabetes (defined as a plasma Hb1Ac ≥ 9.0%)
* Documented history of chronic active inflammatory bowel disorders such as Chrohn's disease or ulcerative colitis
* eGFR of <40 mL/min/1.73 m2 (by Modification of Diet in Renal Disease formula)
* Brachial circumference ≥ 42 cm
* Any history of cerebrovascular event (e.g. stroke, transient ischemic event, cerebrovascular accident)
* Any history of severe cardiovascular event (myocardial infarction, CABG, acute heart failure requiring hospitalization (NYHA III-IV)
* Documented confirmed episode(s) of stable or unstable angina
* Documented repeat (>1) hospitalization for hypertensive crisis within the prior 12 months
* Prescribed to any standard antihypertensive of cardiovascular medication (e.g. beta blockers) for other chronic conditions (e.g. ischemic heart disease) such that discontinuation might pose serious risk to health
* Documented history of persistent or permanent atrial tachyarrhythmia
* Active implantable medical device (e.g. ICD or CRT-D; neuromodulator/spinal stimulator; baroreflex stimulator)
* Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Primary pulmonary hypertension
* Documented contraindication or allergy to contrast medium not amenable to treatment
* Limited life expectancy of < 1 year at the discretion of the Investigator
* Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements or whose participation may result in data analysis confounders (e.g. night shift workers)
* Pregnant, nursing or planning to become pregnant (negative pregnancy test required, documented within a maximum of 7 days prior to procedure for all women of child bearing potential. Documentation of effective contraception is also required for women of child bearing potential) Concurrent enrollment in any other investigational drug or device trial (participation in non-interventional Registries is acceptable)

TRIO Exclusion Criteria

* Renal artery anatomy on either side, ineligible for treatment including:

  * Main renal artery diameter < 3.5 mm and > 8 mm
  * Main renal artery length < 20 mm
  * A single functioning kidney
  * Presence of abnormal kidney tumors
  * Renal artery with aneurysm
  * Pre-existing renal stent or history of renal artery angioplasty
  * Pre-existing aortic stent or history of aortic aneurysm
  * Prior renal denervation procedure
  * Fibromuscular disease of the renal arteries
  * Presence of renal artery stenosis of any origin ≥ 30%
  * Accessory arteries with diameter ≥2 mm <3.5 mm and > 8 mm*
* Iliac/femoral artery stenosis precluding insertion of the Paradise Catheter
* Evidence of active infection within 7 days of procedure
* Secondary hypertension not including sleep apnea (documented through clinical work up within the 12 months prior to consent- see protocol body for details)
* Type I diabetes mellitus or uncontrolled Type II diabetes (defined as a plasma Hb1Ac ≥ 9.0%)
* Documented history of chronic active inflammatory bowel disorders such as Crohn's disease or ulcerative colitis
* eGFR of <40 mL/min/1.73 m2 (by Modification of Diet in Renal Disease formula)
* Brachial circumference ≥ 42 cm
* Any history of cerebrovascular event (e.g. stroke, transient ischemic event, cerebrovascular accident) within 3 months prior to consent
* Any history of severe cardiovascular event (e.g. myocardial infarction, CABG, acute heart failure requiring hospitalization (NYHA III-IV) within 3 months prior to consent
* Documented repeat (>1) hospitalization for hypertensive crisis within the prior 3 months
* Documented confirmed episode(s) of unstable angina within 3 months prior to consent
* Documented intolerance or contraindication for any of the antihypertensive drugs prescribed as a requirement of the study protocol
* Prescribed to any standard anti-hypertensive CV medication (other than beta blockers) for other chronic conditions (e.g. ischemic heart disease) such that discontinuation might pose serious risk to health
* Documented history of persistent or permanent atrial tachyarrhythmia
* Active implantable medical device (e.g. ICD or CRT-D; neuromodulator/spinal stimulator; baroreflex stimulator)
* Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Primary pulmonary hypertension
* Documented contraindication or allergy to contrast medium not amenable to treatment
* Limited life expectancy of < 1 year at the discretion of the Investigator
* Night shift workers
* Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements or whose participation may result in data analysis confounders
* Pregnant, nursing or planning to become pregnant (documented negative pregnancy test required documented within a maximum of 7 days prior to procedure for all women of child bearing potential. Documentation of effective contraception is also required for women of child bearing potential)
* Concurrent enrollment in any other investigational drug or device trial (participation in non-interventional Registries is acceptable)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2025-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Azizi, MD, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou; Ajay J Kirtane, M.D, Principal Investigator — Columbia University
Locations (49):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Health Medical Center, Sacramento, California
  - Stamford Hospital, Stamford, Connecticut
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Southern Illinois University Medicine, Springfield, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ochsner Heart and Vascular Insitute, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Renown Institute for Heart& Vascular Health, Reno, Nevada
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University / NewYork Presbyterian Hospital, New York, New York
  - University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
- Cliniques Universitaires St Luc, Brussels, Belgium
- France (5):
  - Hôpital Saint-André - CHU Bordeaux, Bordeaux
  - CHRU Lille - Institut Coeur Poumon, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Européen Georges-Pompidou, Paris
  - Clinique Pasteur, Toulouse
- Germany (7):
  - University Clinic Dusseldorf, Düsseldorf
  - University Clinic Erlangen, Erlangen
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen GmbH, Freiburg im Breisgau
  - University Clinic of Saarland, Homburg
  - Leipzig Heart Center, Leipzig
  - Sana Kliniken Lübeck GmbH, Lübeck
  - Katholisches Klinikum Mainz, Mainz
- Netherlands (3):
  - Maastricht University Hospital, Maastricht
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Institute of Cardiology, Warsaw
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Imperial College London, Hammersmith Hospital, London, England
  - The Essex Cardiothoracic Centre - Basildon & Thurrock University Hospitals, Basildon
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Conquest Hospital - Hastings, Hastings
  - St Bartholomew's Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Derived] Azizi M, Sharp ASP, Fisher NDL, Weber MA, Lobo MD, Daemen J, Lurz P, Mahfoud F, Schmieder RE, Basile J, Bloch MJ, Saxena M, Wang Y, Sanghvi K, Jenkins JS, Devireddy C, Rader F, Gosse P, Claude L, Augustin DA, McClure CK, Kirtane AJ; RADIANCE Investigators. Patient-Level Pooled Analysis of Endovascular Ultrasound Renal Denervation or a Sham Procedure 6 Months After Medication Escalation: The RADIANCE Clinical Trial Program. Circulation. 2024 Mar 5;149(10):747-759. doi: 10.1161/CIRCULATIONAHA.123.066941. Epub 2023 Oct 26. PMID 37883784
- [Derived] Kirtane AJ, Sharp ASP, Mahfoud F, Fisher NDL, Schmieder RE, Daemen J, Lobo MD, Lurz P, Basile J, Bloch MJ, Weber MA, Saxena M, Wang Y, Sanghvi K, Jenkins JS, Devireddy C, Rader F, Gosse P, Sapoval M, Barman NC, Claude L, Augustin D, Thackeray L, Mullin CM, Azizi M; RADIANCE Investigators and Collaborators. Patient-Level Pooled Analysis of Ultrasound Renal Denervation in the Sham-Controlled RADIANCE II, RADIANCE-HTN SOLO, and RADIANCE-HTN TRIO Trials. JAMA Cardiol. 2023 May 1;8(5):464-473. doi: 10.1001/jamacardio.2023.0338. PMID 36853627
- [Derived] Azizi M, Mahfoud F, Weber MA, Sharp ASP, Schmieder RE, Lurz P, Lobo MD, Fisher NDL, Daemen J, Bloch MJ, Basile J, Sanghvi K, Saxena M, Gosse P, Jenkins JS, Levy T, Persu A, Kably B, Claude L, Reeve-Stoffer H, McClure C, Kirtane AJ; RADIANCE-HTN Investigators. Effects of Renal Denervation vs Sham in Resistant Hypertension After Medication Escalation: Prespecified Analysis at 6 Months of the RADIANCE-HTN TRIO Randomized Clinical Trial. JAMA Cardiol. 2022 Dec 1;7(12):1244-1252. doi: 10.1001/jamacardio.2022.3904. PMID 36350593
- [Derived] Sanghvi K, Wang Y, Daemen J, Mathur A, Jain A, Dohad S, Sapoval M, Azizi M, Mahfoud F, Lurz P, Sayer J, Levy T, Zagoria R, Loening AM, Coleman L, Craig D, Horesh-Bar M, Kirtane AJ. Renal Artery Variations in Patients With Mild-to-Moderate Hypertension From the RADIANCE-HTN SOLO Trial. Cardiovasc Revasc Med. 2022 Jun;39:58-65. doi: 10.1016/j.carrev.2021.09.008. Epub 2021 Sep 30. PMID 34620570
- [Derived] Fisher NDL, Kirtane AJ, Daemen J, Rader F, Lobo MD, Saxena M, Abraham J, Schmieder RE, Sharp ASP, Gosse P, Claude L, Song Y, Azizi M; RADIANCE-HTN Investigators. Plasma renin and aldosterone concentrations related to endovascular ultrasound renal denervation in the RADIANCE-HTN SOLO trial. J Hypertens. 2022 Feb 1;40(2):221-228. doi: 10.1097/HJH.0000000000002994. PMID 34433763
- [Derived] Azizi M, Sanghvi K, Saxena M, Gosse P, Reilly JP, Levy T, Rump LC, Persu A, Basile J, Bloch MJ, Daemen J, Lobo MD, Mahfoud F, Schmieder RE, Sharp ASP, Weber MA, Sapoval M, Fong P, Pathak A, Lantelme P, Hsi D, Bangalore S, Witkowski A, Weil J, Kably B, Barman NC, Reeve-Stoffer H, Coleman L, McClure CK, Kirtane AJ; RADIANCE-HTN investigators. Ultrasound renal denervation for hypertension resistant to a triple medication pill (RADIANCE-HTN TRIO): a randomised, multicentre, single-blind, sham-controlled trial. Lancet. 2021 Jun 26;397(10293):2476-2486. doi: 10.1016/S0140-6736(21)00788-1. Epub 2021 May 16. PMID 34010611
- [Derived] Gosse P, Cremer A, Kirtane AJ, Lobo MD, Saxena M, Daemen J, Wang Y, Stegbauer J, Weber MA, Abraham J, Kario K, Bangalore S, Claude L, Liu Y, Azizi M. Ambulatory Blood Pressure Monitoring to Predict Response to Renal Denervation: A Post Hoc Analysis of the RADIANCE-HTN SOLO Study. Hypertension. 2021 Feb;77(2):529-536. doi: 10.1161/HYPERTENSIONAHA.120.16292. Epub 2020 Dec 28. PMID 33356403
- [Derived] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Lobo MD, Sharp ASP, Bloch MJ, Basile J, Wang Y, Saxena M, Lurz P, Rader F, Sayer J, Fisher NDL, Fouassier D, Barman NC, Reeve-Stoffer H, McClure C, Kirtane AJ; RADIANCE-HTN Investigators. Six-Month Results of Treatment-Blinded Medication Titration for Hypertension Control After Randomization to Endovascular Ultrasound Renal Denervation or a Sham Procedure in the RADIANCE-HTN SOLO Trial. Circulation. 2019 May 28;139(22):2542-2553. doi: 10.1161/CIRCULATIONAHA.119.040451. Epub 2019 Mar 17. PMID 30880441
- [Derived] Calhoun DA, Schiffrin EL, Flack JM. Resistant Hypertension: An Update. Am J Hypertens. 2019 Jan 1;32(1):1-3. doi: 10.1093/ajh/hpy156. No abstract available. PMID 30407514
- [Derived] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590

RESULTS

PARTICIPANT FLOW:
Groups:
- Solo Cohort - Renal Denervation: Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications will be included in the RADIANCE Solo cohort.
  After the post-randomisation qualifying renal angiogram, patients assigned to the renal denervation group underwent immediate endovascular ultrasound nerve ablation with the Paradise endovascular ultrasound renal denervation system.
- Solo Cohort - Sham: Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications will be included in the RADIANCE Solo cohort.
  After the post-randomisation qualifying renal angiogram, patients randomised to the sham group had no further endovascular procedure.
- Trio Cohort - Renal Denervation: Subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications will be included in the RADIANCE Trio cohort.
  After the post-randomisation qualifying renal angiogram, patients assigned to the renal denervation group underwent immediate endovascular ultrasound nerve ablation with the Paradise endovascular ultrasound renal denervation system.
- Trio Cohort - Sham: Subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications will be included in the RADIANCE Trio cohort.
  After the post-randomisation qualifying renal angiogram, patients randomised to the sham group had no further endovascular procedure.
Period: Overall Study
Arm/Group | Solo Cohort - Renal Denervation | Solo Cohort - Sham | Trio Cohort - Renal Denervation | Trio Cohort - Sham
Started | 74 | 72 | 69 | 67
Patient Crossed-over From Sham to Renal Denervation | 0 | 37 | 0 | 22
Completed | 73 | 46 | 41 | 36
Not Completed | 1 | 26 | 28 | 31
Not completed — Follow-up on going | 1 | 26 | 28 | 31

BASELINE CHARACTERISTICS:
Groups:
- Solo Cohort - Renal Denervation; Solo Cohort - Sham: Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications will be included in the RADIANCE Solo cohort
- Trio Cohort - Renal Denervation; Trio Cohort - Sham: Subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications will be included in the RADIANCE Trio cohort.
- Total: Total of all reporting groups
Arm/Group | Solo Cohort - Renal Denervation | Solo Cohort - Sham | Trio Cohort - Renal Denervation | Trio Cohort - Sham | Total
Number analyzed (Participants) | 74 | 72 | 69 | 67 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 74 | 72 | 69 | 67 | 282
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.2) | 53.8 (10.0) | 52.3 (7.5) | 52.8 (9.1) | 53.32 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 13 | 14 | 88
  Male | 46 | 39 | 56 | 53 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 60 | 52 | 44 | 50 | 206
  Black | 12 | 13 | 14 | 13 | 52
  Other or unknown | 2 | 7 | 11 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Solo Cohort - Mean Difference in Average Daytime Ambulatory Systolic BP
Description: Mean difference in average daytime ambulatory systolic BP of the Solo cohort
Time Frame: from baseline to 2 months post procedure
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Solo Cohort - Renal Denervation | Solo Cohort - Sham
Number analyzed (Participants) | 74 | 72
mm Hg | -8.5 (9.3) | -2.2 (10.0)

2. Secondary Outcome: Reduction in Average 24-hr/Night-time Ambulatory Systolic BP
Time Frame: from baseline to 2 months post procedure
Reporting Status: Not Posted

3. Secondary Outcome: Reduction in Average Daytime/24-hr/Night-time Diastolic BP
Time Frame: from baseline to 2 months post procedure
Reporting Status: Not Posted

4. Secondary Outcome: All-cause Mortality
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

5. Secondary Outcome: Hypertensive or Hypotensive Emergency Resulting in Hospitalization
Time Frame: up to 36 months
Reporting Status: Not Posted

6. Secondary Outcome: Hospitalization for Heart Failure
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

7. Secondary Outcome: Stroke, Transient Ischemic Attack, Cerebrovascular Accident
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

8. Secondary Outcome: Acute Myocardial Infarction
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

9. Secondary Outcome: End Stage Renal Disease
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

10. Secondary Outcome: Renal Artery or Vascular Complications Requiring Intervention
Time Frame: from baseline to 36 months post-procedure
Reporting Status: Not Posted

11. Secondary Outcome: Significant Embolic Events Resulting in End Organ Damage
Time Frame: from baseline to 1 month and 36 months post-procedure
Reporting Status: Not Posted

12. Secondary Outcome: Procedure Related Pain Lasting > 2 Days
Time Frame: from baseline to 1 month and 36 months post-procedure
Reporting Status: Not Posted

13. Secondary Outcome: Acute Renal Injury
Time Frame: from baseline to 1 month and 36 months post-procedure
Reporting Status: Not Posted

14. Secondary Outcome: Significant (>50%) and Severe (>75%) New Onset Renal Stenosis
Description: as diagnosed by duplex ultrasound and confirmed by renal CTA/MRA or as diagnosed/confirmed by study defined renal CTA/MRA at 12 months
Time Frame: from baseline to 6, 12, 24 and 36 months post-procedure
Reporting Status: Not Posted

15. Secondary Outcome: Major Access Site Complications
Time Frame: from baseline to 1 month and 36 months post-procedure
Reporting Status: Not Posted

16. Primary Outcome: Trio Cohort - Median Change in Daytime Ambulatory Systolic BP
Description: Median change in daytime ambulatory systolic BP of the Trio cohort
Time Frame: from baseline to 2 months post procedure
Population: Intention-to-treat population
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Trio Cohort - Renal Denervation | Trio Cohort - Sham
Number analyzed (Participants) | 69 | 67
mm Hg | -8 [-16.4 to 0] | -3 [-10.3 to 1.8]

ADVERSE EVENTS:
Time Frame: List of AE and SAE by term and by arm at 2 months post-procedure (0-67 days post-procedure)
Description: For the cross-over group, AEs were collected and we reported here the list of AE and SAE over the period of 0 to 67 days post-cross-over procedure.
Groups:
- Solo Cohort - Treatment Group: Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications were included in the RADIANCE Solo cohort and were treated by renal denervation
- Solo Cohort - Sham Group: Subjects with essential hypertension controlled on 1 or 2 antihypertensive medications or uncontrolled on 0-2 antihypertensive medications were included in the RADIANCE Solo cohort with the option for cross-over treatment after 6-months
- Trio Cohort - Treatment Group: Subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications were included in the RADIANCE Trio cohort, were treated by renal denervation with maintenance of anti-hypertensive medications
- Trio Cohort - Sham Group: Subjects with treatment resistant hypertension on a minimum of 3 antihypertensive medications were included in the RADIANCE Trio cohort were maintained with anti-hypertensive medications with option for cross-over treatment after 6-months
- Cross-over Group: Subjects from Solo and Trio cohorts who crossed over to the treatment arm after 6-months post-randomization.
Arm/Group | Solo Cohort - Treatment Group | Solo Cohort - Sham Group | Trio Cohort - Treatment Group | Trio Cohort - Sham Group | Cross-over Group
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/72 | 1/69 | 0/67 | 1/59
Serious Adverse Events (participants affected / at risk) | 7/74 | 0/72 | 12/69 | 4/67 | 1/59
Other Adverse Events (participants affected / at risk) | 60/74 | 40/72 | 56/69 | 34/67 | 19/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solo Cohort - Treatment Group (N=74) | Solo Cohort - Sham Group (N=72) | Trio Cohort - Treatment Group (N=69) | Trio Cohort - Sham Group (N=67) | Cross-over Group (N=59)
Atrioventricular block - Drug therapy (Cardiac disorders) | 1 (1) | 0 (0) | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 | 0 | 0
Bradycardia - Drug therapy (Cardiac disorders) | 2 (2) | 0 (0) | 0 | 0 | 0
Hematoma Infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Hypotension (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 2 (3) | 0 | 0
Presyncope - Drug therapy (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0
Sedation complication - Drug therapy (Surgical and medical procedures) | 0 | 0 | 1 (1) | 0 | 0
Vascular access site haematoma (Surgical and medical procedures) | 0 | 0 | 1 (1) | 0 | 0
Vascular pseudoaneurysm (Surgical and medical procedures) | 0 | 0 | 1 (1) | 0 | 0
Adverse drug reaction - Sevikar HCT (Amlodipine, Olmesartan and Hydrochlorothiazide) (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0
Blood sodium abnormal (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 (1) | 0
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 0 | 0 | 1 (1) | 0
Death (General disorders) | 0 | 0 | 1 (1) | 0 | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 (2) | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 — Independent review of preprocedural and 6-month post procedure renal artery imaging showed that there was a pre-existing ostial renal artery stenosis which would have met the criteria for exclusion but was not recognized at the time of randomization.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solo Cohort - Treatment Group (N=74) | Solo Cohort - Sham Group (N=72) | Trio Cohort - Treatment Group (N=69) | Trio Cohort - Sham Group (N=67) | Cross-over Group (N=59)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 5 (5) | 6 (6) | 6 (6)
Vascular access site haematoma (Surgical and medical procedures) | 11 (11) | 13 (13) | 10 (10) | 5 (5) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 5 (6)
Vascular access site pain (Surgical and medical procedures) | 13 (13) | 10 (10) | 9 (9) | 9 (9) | 5 (5)
Vasospasm (Vascular disorders) | 15 (15) | 0 (0) | 13 (13) | 1 (1) | 3 (3)
Headache (General disorders) | 5 (5) | 6 (7) | 3 (5) | 5 (5) | 0 (0)
Hypertension - Condition aggravated (Cardiac disorders) | 3 (3) | 9 (9) | 2 (2) | 7 (8) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Vasospasm - Drug therapy (Vascular disorders) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02649426/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02649426/SAP_001.pdf